CLINICAL TRIAL: NCT06454773
Title: To Evaluate the Impact of Consumption of Bioactive Compounds Extracted From Hemp Hull and Black Pepper on Fasting Blood Glucose Levels in People With Pre-diabetes: A Randomized Placebo-Controlled Parallel Arm Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Collaborators: Brightseed (Industry)
Responsible Party: Principal Investigator, Dr Anoop Misra, Professor, President, Diabetes Foundation, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: F.No 1.4 FCDOC/EC/HAO/2024-25
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Intervention

STUDY DESIGN:
Intervention Model Description: double-blind placebo controlled
Who Masked: Participant, Investigator
Masking Description: Bioactive extract vs placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): bioactive compound from black pepper and hemp hull
  Interventions: Dietary Supplement: NCT/NFT
- control (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: NCT/NFT

INTERVENTIONS:
Dietary Supplement: NCT/NFT — extract from black pepper and hemp hull

SUMMARY:
This is randomized controlled parallel arm study on free living Asian Indians. Eligible subjects will undergo one-week run-in period and subjects will be asked to maintain their usual diet and exercise regime. At the end of the run-in period, subjects fulfilling the inclusion/exclusion criteria at this stage will be randomized either to the intervention arm or control arm using computerized random number tables.

The measured parameters will include, 24-h diet recall, food frequency questionnaire, anthropometry including circumferences, height and weight, and blood parameters including blood glucose (fasting), serum insulin (fasting), HbA1c and lipid profile.

DETAILED DESCRIPTION:
To study the impact of bioactive compound supplementation on fasting blood glucose.

To study the impact of intervention with bioactive compound on following measures of glycaemia:

* 24 hr AUC total from CGM Post-prandial glucose regulation
* iAUC determined from CGM readout up to 2 hr after consumption of a Standard Meal Blood Chemistry
* Fasting Insulin
* HbA1c
* Lipid profile Anthropometry
* Weight
* BMI
* Waist Circumference

ELIGIBILITY:
Inclusion Criteria:

* Prediabetic individuals of BMI range 25-30 kg/m2 and waist circumference ≥80cm for women and ≥90cm for men with Fasting Blood Glucose between 100-125 mg/dL.

Exclusion Criteria:

* Prediabetic individuals of BMI range 25-30 kg/m2 and waist circumference ≥80cm for women and ≥90cm for men with Fasting Blood Glucose between 100-125 mg/dL.

Exclusion criteria

1. Weight loss or gain ≥4.5 kg within 90 days of visit 1.
2. Use of weight loss medications within 90 days of visit 1
3. History of gastrointestinal surgery (e.g., bariatric surgery) or cosmetic procedures (e.g., liposuction) for weight/fat reducing purposes.
4. Use of dietary supplements or related products that, in the judgment of the Investigator, are likely to markedly affect weight loss or appetite within 30 days of visit 1.
5. History of extreme dietary habits (e.g., Atkins diet, etc.), as judged by the Investigator.
6. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
7. Current medical diagnosis of type 1 or type 2 diabetes mellitus.
8. HbA1c ≥48 mmol/mol (6.5%) as measured at visit 1.
9. History of a chronic gastrointestinal disorder, such as peptic ulcer disease or malabsorption syndrome (mild lactose intolerance or gastroesophageal reflux diseases are acceptable).
10. Signs or symptoms of an active infection of clinical relevance within 5 days of visit 1. The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to visit 1.
11. Is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source document.
12. Any condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.
13. Excessive alcohol consumption (> 2 Drinks, 60 ml of Whisky Per Day).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
fasting blood glucose | 30 days

SECONDARY OUTCOMES:
Body weight | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Diabetes, obesity and cholesterol foundation (NDOC), Delhi, India